CLINICAL TRIAL: NCT01522911
Title: Interventional Study to Investigate the Effects of Percutaneous Closure of the Left Atrial Appendage on Atrial and Brain Natriuretic Peptide Secretion
Brief Title: Atrial and Brain Natriuretic Peptide Secretion After Percutaneous Closure of the Left Atrial Appendage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Nicolas Majunke, senior physician, University of Leipzig
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAA-1
Record Dates: First submitted 2011-12-20; First posted 2012-02-01 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Atrial Fibrillation; Stroke Prevention; Left Atrial Appendage
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- atrial and brain natriuretic peptide (Other): Impact on atrial an brain natriuretic peptide secretion after percutaneous left atrial appendage closure
  Interventions: Device: WATCHMAN LAA system (Percutaneous left atrial appendage closure)

INTERVENTIONS:
Device: WATCHMAN LAA system (Percutaneous left atrial appendage closure) — The WATCHMAN LAA system (Altritech Inc., Plymouth, MN),Percutaneous occlusion systems have been developed as an alternative to anticoagulation for stroke prevention. Briefly, transseptal puncture is performed to gain access to the left atrial appendage (LAA). Thereafter LAA angiography is performed. After an optimal device size is chosen based on LAA measurements by fluoro and echocardiography the occluder is implanted into the orifice of the left atrial appendage under fluoroscopy and TEE-guidance. The size of the device is chosen to be 10% to 20% larger than diameter of the LAA ostium to have stable positioning of the device. Every procedure is performed under local anaesthesia. Heparin is given during implantation procedure to achieve an activated clotting time of at least 250.

SUMMARY:
To date there are no data suggesting substantial effects of hormonal interaction after percutaneous closure of the left atrial appendage (LAA). Our hypothesis is that by excluding the LAA from blood flow physiologic stimuli for ANP and BNP produce may be impaired and consecutive release of the hormones may be reduced. Here, we present our experience of ANP and BNP secretion in the early postprocedural period after transcatheter closure of the LAA.

ELIGIBILITY:
Inclusion Criteria:

* non-valvular atrial fibrillation
* increased risk for thromboembolic complications (a minimum CHADS2Score of at least 2)

Exclusion Criteria:

* Valvular-atrial fibrillation
* Low risk for thromboembolic complications CHADS-2-Score < 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-05; Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Plasma ANP and BNP levels after transcatheter closure of the left atrial appendage. | participants will be followed for the duration of hospital stay, an expected average of 48 hours
  Venous blood samples are taken before the procedure, immediately after implantation of the LAA closure device and on the first morning after the procedure. The blood is drawn into plastic tubes containing aprotinin and ethylenediaminetetraacetic acid disodium and is promptly centrifuged. The plasma obtained is stored at -20°C until assayed. The plasma BNP and ANP concentrations are then determined with a commercially available enzyme immunoassay kit (ELISA Kit for Brain Natriuretic Peptide, Uscn Life Science Inc., Missouri City, USA and ANP ELISA Kit, Hölzel Diagnostika, Köln, Germany).

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Majunke, M.D., Principal Investigator — HearCenter Leipzig; Sven Moebius-Winkler, M.D., Principal Investigator — HearCenter Leipzig; Gerhard Schuler, Professor, Principal Investigator — HearCenter Leipzig